CLINICAL TRIAL: NCT00087529
Title: A Phase II/III, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Multicenter Study to Evaluate the Safety and Efficacy of Rituximab in Adults With Primary Progressive Multiple Sclerosis
Brief Title: A Study to Evaluate the Safety and Efficacy of Rituximab in Adults With Primary Progressive Multiple Sclerosis
Acronym: OLYMPUS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Clinical Trials Posting Group, Genentech, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U2786g
Record Dates: First submitted 2004-07-09; First posted 2004-07-13 (Estimated); Results first posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-08

CONDITIONS: Multiple Sclerosis
Keywords: PPMS; Primary progressive MS; Primary progressive multiple sclerosis; Rituxan; MS
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Chronic Progressive | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: rituximab
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: placebo — Intravenous repeating dose
  Arms: 2
Drug: rituximab — Intravenous repeating dose
  Arms: 1

SUMMARY:
This is a Phase II/III, randomized, double-blind, parallel group, placebo controlled, multicenter study to evaluate the safety and efficacy of rituximab in adults with PPMS. The study will enroll approximately 435 subjects at up to 60 sites in the United States and Canada.

ELIGIBILITY:
Inclusion Criteria:

* Definitive diagnosis of PPMS
* Disease duration of ≥ 1 year
* EDSS at baseline between 2.0 and 6.5 points, inclusive
* Score of ≥ 2.0 on the Functional Systems (FS) scale for the pyramidal system or gait that is due to lower extremity findings
* Presence of at least one of the following in a CSF specimen obtained during the screening period and analyzed by the central laboratory or results from a CSF sample obtained during the previous 24 months:
* For subjects of reproductive potential (males and females), use of a reliable means of contraception (e.g., hormonal contraceptive, patch, vaginal ring, intrauterine device, physical barrier) during study treatment and for 1 year following the last dose of study drug

Exclusion Criteria:

* Pregnancy or lactation
* Incompatibility with MRI
* Lack of peripheral venous access
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Known active bacterial, viral, fungal, mycobacterial, or other infection (including atypical mycobacterial disease, but excluding fungal infections of nail beds or recurrent herpes zoster or simplex infections) or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 30 days prior to screening or oral antibiotics within 14 days prior to screening
* History or presence of recurrent or chronic infection (e.g., hepatitis B or C, HIV, syphilis)
* History of cancer, including solid tumors and hematologic malignancies (except resected and fully resolved cutaneous basal cell and squamous cell carcinomas)
* History of alcohol or drug abuse within 6 months prior to screening
* History of or currently active primary or secondary immunodeficiency
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease)
* Presence of other significant, uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, or gastrointestinal disease that might interfere with a subject's ability to participate and to complete approximately 2.5 years of study participation
* History or presence of MS relapse or exacerbation
* History or presence of vascular disease potentially affecting the brain or spinal cord (e.g., stroke, transient ischemic attack, carotid stenosis, aortic aneurysm, intracranial aneurysm, hemorrhage, arteriovenous malformation)
* History or presence of myelopathy due to spinal cord compression by disk or vertebral disease
* History of severe, clinically significant central nervous system trauma (e.g., cerebral contusion, spinal cord compression)
* History of intracranial or intraspinal tumor (e.g., meningioma, glioma)
* History or presence of potential metabolic cause of myelopathy or encephalopathy (e.g., vitamin B12 deficiency, thyroid abnormalities)
* History or presence of infectious causes of myelopathy (e.g., syphilis, Lyme disease, human T-cell lymphotropic virus type 1 [HTLV-1], or herpes zoster myelopathy)
* History of genetically inherited progressive CNS degenerative disorder (e.g., X-linked adrenoleukodystrophy, hereditary spastic paraparesis)
* Neuromyelitis optica
* History or presence of systemic autoimmune disorders potentially causing progressive neurologic disease (e.g., lupus, anti-phospholipid antibody syndrome, Sj�gren syndrome, Beh�et disease)
* History or presence of sarcoidosis
* Previous treatment with rituximab (MabThera(R)/Rituxan(R))
* Previous treatment with lymphocyte-depleting therapies (e.g., cyclophosphamide, Campath(R), anti-CD4, cladribine, total body irradiation, bone marrow transplantation), except mitoxantrone, which should not be used 12 months prior to randomization
* Treatment with an investigational agent within 90 days or 5 half-lives of the investigational drug (whichever is longer) prior to randomization
* Receipt of a live vaccine within 30 days prior to randomization
* Systemic corticosteroid therapy within 30 days prior to randomization
* Treatment with IFN-β, glatiramer acetate, IVIg, or plasmapheresis within 60 days prior to randomization
* Treatment with non-lymphocyte-depleting immunosuppressive therapies (e.g., azathioprine, mycophenolate mofetil [MMF], cyclosporine) within 90 days prior to randomization
* Statins or hormone replacement therapy started within 30 days prior to randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2004-06; Primary Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Smith, M.D., Study Director — Genentech, Inc.

REFERENCES:
- [Derived] Kappos L, Yiu S, Dahlke F, Coetzee T, Cutter GR, Yuen S, Bonati U, Lublin FD. Composite Confirmed Disability Worsening/Progression Is a Useful Clinical Endpoint for Multiple Sclerosis Clinical Trials. Neurology. 2025 May 27;104(10):e213558. doi: 10.1212/WNL.0000000000213558. Epub 2025 Apr 21. PMID 40258203
- [Derived] Falet JR, Durso-Finley J, Nichyporuk B, Schroeter J, Bovis F, Sormani MP, Precup D, Arbel T, Arnold DL. Estimating individual treatment effect on disability progression in multiple sclerosis using deep learning. Nat Commun. 2022 Sep 26;13(1):5645. doi: 10.1038/s41467-022-33269-x. PMID 36163349
- [Derived] Zhang J, Waubant E, Cutter G, Wolinsky JS, Glanzman R. EDSS variability before randomization may limit treatment discovery in primary progressive MS. Mult Scler. 2013 May;19(6):775-81. doi: 10.1177/1352458512459685. Epub 2012 Oct 1. PMID 23027880
- [Derived] Hawker K, O'Connor P, Freedman MS, Calabresi PA, Antel J, Simon J, Hauser S, Waubant E, Vollmer T, Panitch H, Zhang J, Chin P, Smith CH; OLYMPUS trial group. Rituximab in patients with primary progressive multiple sclerosis: results of a randomized double-blind placebo-controlled multicenter trial. Ann Neurol. 2009 Oct;66(4):460-71. doi: 10.1002/ana.21867. PMID 19847908

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received the placebo equivalent to rituximab via IV infusion, for a treatment period of 96 weeks. Each treatment course involved 2 separate infusions of placebo separated by 14 days without study drug. The first course was administered on Days 1 and 15, and subsequent courses were initiated every 24 weeks.
- Rituximab: Participants received rituximab 1 gram via IV infusion, for a treatment period of 96 weeks. Each treatment course involved 2 separate infusions of rituximab separated by 14 days without study drug. The first course was administered on Days 1 and 15, and subsequent courses were initiated every 24 weeks.
Period: Overall Study
Arm/Group | Placebo | Rituximab
Started | 147 | 292
Completed | 116 | 224
Not Completed | 31 | 68
Not completed — Death | 1 | 0
Not completed — Adverse Event | 0 | 8
Not completed — Pregnancy | 0 | 1
Not completed — Lost to Follow-up | 2 | 3
Not completed — Participant Decision | 14 | 37
Not completed — Physician Decision | 4 | 8
Not completed — Initiation of Excluded Therapy | 0 | 1
Not completed — Participant Noncompliance | 0 | 1
Not completed — Disease Progression | 5 | 4
Not completed — Did Not Continue to Safety Follow-Up | 5 | 5

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All randomized participants, with groups defined by treatment assigned at randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rituximab | Total
Number analyzed (Participants) | 147 | 292 | 439
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (8.69) | 50.1 (9.02) | 49.9 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 140 | 221
  Male | 66 | 152 | 218

OUTCOME MEASURES:

1. Primary Outcome: Time to Confirmed Disease Progression (CDP)
Description: Disease progression was assessed using the Expanded Disability Status Scale (EDSS), a disability scale that ranges from 0 to 10, where higher scores represent increased disability. Progression was defined as either an increase of greater than or equal to (≥) 1 point from a Baseline EDSS score within 2.0 to 5.5 points, or an increase of ≥0.5 points from a Baseline EDSS score greater than (>) 5.5 points, for which the change was not attributable to another etiology. Repeat assessment to determine CDP must have occurred at a regularly scheduled visit at least 12 weeks after initial progression; those who discontinued treatment early without confirmatory EDSS assessment were considered as having CDP. Those who did not meet criteria for CDP, completed treatment with only initial progression, or received an exclusionary therapy were censored at last EDSS assessment. Time to CDP was the time from randomization to initial disease progression, estimated using Kaplan-Meier (KM) analysis.
Time Frame: 96 weeks (from Screening to Week 96, and at least 12 weeks after initial progression)
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 147 | 292
weeks | NA [NA to NA] — Stratified log rank test was used to test treatment effect. Hazard ratio and CDP rate (from KM) were used to describe treatment effect. Median time to CDP was not available because less than (<) 50 percent (%) had a CDP event by end of Week 96. | NA [NA to NA] — Stratified log rank test was used to test treatment effect. Hazard ratio and CDP rate (from KM) were used to describe treatment effect. Median time to CDP was not available because less than (<) 50 percent (%) had a CDP event by end of Week 96.
Statistical Analysis 1: Comparison: Placebo vs Rituximab; Test type: Superiority or Other; p = 0.1442, Log Rank — Stratified using the following variables: Baseline EDSS (less than or equal to [≤] 4.0 versus >4.0 points) and prior treatment with interferon-beta or glatiramer acetate; Hazard Ratio (HR) = 0.773, 95% CI 2-sided [0.546 to 1.093]

2. Primary Outcome: Percentage of Participants With CDP
Description: Disease progression was assessed using the EDSS, a disability scale that ranges from 0 to 10, where higher scores represent increased disability. Progression was defined as either an increase of ≥1 point from a Baseline EDSS score within 2.0 to 5.5 points, or an increase of ≥0.5 points from a Baseline EDSS score >5.5 points, for which the change was not attributable to another etiology. Repeat assessment to determine CDP must have occurred at a regularly scheduled visit at least 12 weeks after initial progression; those who discontinued treatment early without confirmatory EDSS assessment were considered as having CDP. The percentage of participants with CDP was calculated as [number of participants meeting the above criteria divided by the number analyzed] multiplied by 100.
Time Frame: 96 weeks (from Screening to Week 96, and at least 12 weeks after initial progression)
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 147 | 292
percentage of participants | 36.1 | 28.4

3. Secondary Outcome: Change From Baseline to Week 96 in Total Volume of Transverse Relaxation Time (T2) Brain Lesions on Magnetic Resonance Imaging (MRI) Scan
Description: Scheduled T2-weighted MRI scans of the brain and cervical spinal cord were performed with and without gadolinium contrast at Screening and Week 6, and without gadolinium at Weeks 48, 96, and 122 and/or upon early termination. The total volume of T2 (ie, hyperintense) brain lesions at each visit was documented. Missing Week 96 values were imputed using a last observation carried forward (LOCF) approach, while participants with missing Baseline values were excluded. The change in T2 lesion volume was calculated as [volume at Week 96 minus volume at Baseline] and expressed in cubic millimeters (mm^3).
Time Frame: At Baseline and Week 96
Population: ITT Population. Participants with missing Baseline values were excluded.
Measure: Median (Full Range); unit: mm^3
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 147 | 290
mm^3 | 809.50 [-8557.00 to 26367.00] | 301.95 [-4031.00 to 24076.00]
Statistical Analysis 1: Comparison: Placebo vs Rituximab; Treatment difference in least-squares (LS) means and the associated 95% confidence intervals were estimated from the analysis of variance (ANOVA) model, which included the following factors: Baseline EDSS (≤ 4.0 versus >4.0 points), prior treatment with interferon-beta or glatiramer acetate, and treatment group; Test type: Superiority or Other; p = 0.0008, Friedman ranked ANOVA test; LS mean difference = -718.24, 95% CI 2-sided [-1504.48 to 68.00]

4. Secondary Outcome: Change From Baseline to Week 96 in Brain Volume on MRI Scan
Description: Scheduled MRI scans of the brain and cervical spinal cord were performed with and without gadolinium contrast at Screening and Week 6, and without gadolinium at Weeks 48, 96, and 122 and/or upon early termination. The total brain volume was documented at Baseline and at visits occurring during Weeks 48 and 96. Missing Week 96 values were imputed using a LOCF approach, while participants with missing Baseline values were excluded. The change in brain volume was calculated as [volume at Week 96 minus volume at Baseline] and expressed in cubic centimeters (cm^3).
Time Frame: At Baseline and Week 96
Population: ITT Population. Participants with missing Baseline values were excluded.
Measure: Median (Full Range); unit: cm^3
Arm/Group | Placebo | Rituximab
Number analyzed (Participants) | 130 | 237
cm^3 | -14.00 [-76.00 to 323.70] | -13.10 [-91.00 to 346.40]
Statistical Analysis 1: Comparison: Placebo vs Rituximab; Treatment difference in LS means and the associated 95% confidence intervals were estimated from the ANOVA model, which included the following factors: Baseline EDSS (≤ 4.0 versus >4.0 points), prior treatment with interferon-beta or glatiramer acetate, and treatment group; Test type: Superiority or Other; p = 0.6237, Friedman ranked ANOVA test; LS mean difference = -1.08, 95% CI 2-sided [-9.49 to 7.34]

ADVERSE EVENTS:
Time Frame: Up to 122 weeks (from start of first infusion until study completion or early termination)
Arm/Group | Placebo | Rituximab
Serious Adverse Events (participants affected / at risk) | 20/147 | 47/292
Other Adverse Events (participants affected / at risk) | 147/147 | 289/292
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=147) | Rituximab (N=292)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 2
Myocardial infarction (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Appendicitis perforated (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 1
Abasia (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 4
Bronchitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Heart rate irregular (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 4
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Cerebellar ataxia (Nervous system disorders) | 0 | 1
Multiple sclerosis (Nervous system disorders) | 1 | 1
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0
Myelitis transverse (Nervous system disorders) | 0 | 1
Muscle spasticity (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 1 | 0
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Activities of daily living impaired (Social circumstances) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=147) | Rituximab (N=292)
Vision blurred (Eye disorders) | 9 | 15
Nausea (Gastrointestinal disorders) | 16 | 55
Constipation (Gastrointestinal disorders) | 20 | 29
Diarrhoea (Gastrointestinal disorders) | 13 | 23
Vomiting (Gastrointestinal disorders) | 10 | 17
Dyspepsia (Gastrointestinal disorders) | 2 | 15
Fatigue (General disorders) | 46 | 104
Gait disturbance (General disorders) | 34 | 60
Oedema peripheral (General disorders) | 15 | 45
Asthenia (General disorders) | 17 | 36
Pyrexia (General disorders) | 9 | 39
Chills (General disorders) | 6 | 35
Pain (General disorders) | 8 | 21
Influenza like illness (General disorders) | 3 | 16
Chest pain (General disorders) | 8 | 8
Urinary tract infection (Infections and infestations) | 36 | 68
Nasopharyngitis (Infections and infestations) | 38 | 64
Upper respiratory tract infection (Infections and infestations) | 27 | 45
Influenza (Infections and infestations) | 9 | 22
Sinusitis (Infections and infestations) | 9 | 19
Bronchitis (Infections and infestations) | 3 | 15
Fall (Injury, poisoning and procedural complications) | 40 | 96
Contusion (Injury, poisoning and procedural complications) | 19 | 41
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 18 | 37
Procedural pain (Injury, poisoning and procedural complications) | 11 | 18
Excoriation (Injury, poisoning and procedural complications) | 6 | 20
Muscular weakness (Musculoskeletal and connective tissue disorders) | 42 | 101
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 66
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 59
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 | 56
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 17 | 44
Muscle spasms (Musculoskeletal and connective tissue disorders) | 22 | 37
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 29
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 23
Neck pain (Musculoskeletal and connective tissue disorders) | 8 | 22
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 17
Headache (Nervous system disorders) | 27 | 77
Hypoaesthesia (Nervous system disorders) | 32 | 57
Muscle spasticity (Nervous system disorders) | 32 | 49
Paraesthesia (Nervous system disorders) | 19 | 41
Dizziness (Nervous system disorders) | 15 | 42
Balance disorder (Nervous system disorders) | 21 | 31
Tremor (Nervous system disorders) | 12 | 20
Burning sensation (Nervous system disorders) | 7 | 20
Ataxia (Nervous system disorders) | 6 | 18
Depression (Psychiatric disorders) | 25 | 34
Insomnia (Psychiatric disorders) | 12 | 40
Anxiety (Psychiatric disorders) | 7 | 15
Micturition urgency (Renal and urinary disorders) | 10 | 21
Pollakiuria (Renal and urinary disorders) | 8 | 11
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 15 | 34
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 33
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 24
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 22
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 17
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 64
Rash (Skin and subcutaneous tissue disorders) | 13 | 49
Erythema (Skin and subcutaneous tissue disorders) | 3 | 21
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 17
Flushing (Vascular disorders) | 7 | 39
Hypotension (Vascular disorders) | 12 | 30
Hypertension (Vascular disorders) | 10 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.